CLINICAL TRIAL: NCT05647746
Title: Performance Comparison of Compumedics Somfit Sleep Monitoring Device Against Home Sleep Apnoea Testing Device (Itamar WatchPAT) and Polysomnography
Brief Title: Comparative Assessment of Compumedics Somfit Sleep Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Compumedics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AJ259
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: As the study investigate performances of the diagnostic equipment, the three diagnostic devices can be applied to the single group of patients at the same time
Who Masked: Outcomes Assessor
Masking Description: The sleep technologists who assess the sleep study outcomes will be blinded to the device generating the diagnostic data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Compumedics Somfit HSAT device, WatchPAT HSAT device, Compumedics Grael /E-series PSG system — Each intervention is a separate diagnostic device. They will all be operating at the same time

SUMMARY:
To study whether Somfit is substantially equivalent to the existing approved devices for full polysomnography and home sleep apnea testing

DETAILED DESCRIPTION:
Sleep is recognized as one of the three pillars of health (i.e. nutrition, exercise and sleep). Poor quality and fragmented sleep leads to an increase in the risk for development of chronic health conditions. Given the importance of good quality sleep and its critical role in overall well-being, there is a need for regular monitoring and assessment of sleep quality in individuals. However, current technologies will only allow for this to be performed in sleep clinics and with the help of full polysomnography (PSG) systems which require the patients to spend a night at the clinic with several wired electrodes connected to their scalp. This "gold standard" technology is expensive and therefore does not allow to meet public health demand for diagnosis of sleep disorders, especially obstructive sleep apnea (OSA) and also can be uncomfortable for the patients and distort their natural sleep architecture. To solve this problem, Compumedics has recently developed a miniaturized, portable, automated and affordable sleep monitoring system with code name of "Somfit" which is attached to patients' forehead and can be used in the comfort of patients' home. While Somfit has already gained TGA approval, the aim of this study is to compare Somfit with the "gold standard" PSG and another approved portable sleep testing device, Itamar WatchPAT One, in terms of accuracy of characterising sleep neurological architecture and diagnosing OSA, with the objective of applying for the international regulatory approvals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or over
* Be able to give informed consent
* Referral for a diagnostic sleep study with indication of suspected sleep disordered breathing or history of diagnosed sleep disordered breathing

Exclusion Criteria:

* Less than 18 years of age
* Unable or not willing to provide informed consent
* Need for nursing attendance during the time between 9 pm and 9 am
* Use of any OSA treatments during any part of the PSG study
* Previous reaction to skin preparation, tapes and electrode gels used at PSG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The AHI difference between the test device (Somfit) and gold standard (PSG) | Data required for the primary outcome measure are generated in the course of single night sleep recording for every participant. Statistical estimation will be performed after completion of all sleep recordings
  AHI is the apnea hypopnea index, main measure of presence/severity of OSA (obstructive sleep apnea). it will test the null hypothesis that Somfit AHI is not equivalent to the AHI reported by PSG
The AHI difference between the test device (Somfit) and predicate device (WatchPAT) | Data required for this primary outcome measure are generated in the course of single night sleep recording for every participant. Statistical estimation will be performed after completion of all sleep recordings
  AHI is the apnea hypopnea index, main measure of presence/severity of OSA (obstructive sleep apnea). it will test the null hypothesis that Somfit AHI is not equivalent to the AHI reported by PSG

SECONDARY OUTCOMES:
Difference between hypnogram percent agreements between WatchPAT and PSG, and between Somfit and PSG | Data required for this outcome measure are generated in the course of single night sleep recording for every participant. Statistical estimation will be performed after completion of all sleep recordings
  It will test the null hypothesis that the accuracy of sleep staging performed by the test device (Somfit) is inferior to that of the predicate device (WatchPAT)
Hypnogram percent agreement between Somfit and PSG | Data required for this outcome measure are generated in the course of single night sleep recording for every participant. Statistical estimation will be performed after completion of all sleep recordings
  It will test the null hypothesis that the accuracy of sleep staging performed by the test device (Somfit) is inferior to that demonstrated by the accredited sleep technologists

OTHER OUTCOMES:
Respiratory Event Index (REI) for Somfit | The measure will be calculated for every participant following a single night sleep recording
  Additional outcome for sleep quality
Oxygen Desaturation Index (ODI) for Somfit | The measure will be calculated for every participant following a single night sleep recording
  Additional outcome for sleep quality
Average pulse rate (PR) for Somfit | The measure will be calculated for every participant following a single night sleep recording
  Additional outcome for sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- SleepMetrics Pty Ltd, Heidelberg, VUC, Australia

IPD SHARING:
Plan to Share IPD: No